CLINICAL TRIAL: NCT06050382
Title: Investigation Of The Effect Of Progressive Relaxation Training On Pain Characteristics, Attack Frequency, Perception Of Activity Self-Efficiency And Social Participation In Women With Tension-Type Headache And Migraine
Brief Title: Progressive Relaxation Training Effect On Pain, Activity And Social Participation In Women With Tension-Type Headache And Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gokcen Akyurek, Assoc Prof, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08.11.2022/3
Record Dates: First submitted 2023-08-18; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Pain, Chronic; Migraine Disorders; Tension-Type Headache
Keywords: pain; women; progressive relaxation training; participation
MeSH Terms: conditions — Chronic Pain; Migraine Disorders; Tension-Type Headache; Pain | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WOMEN WITH TENSION-TYPE HEADACHE (Experimental): The tension headache group consists of 22 women aged 20-45 years.The inclusion criteria were determined as follows being between the ages of 20 and 45, having a diagnosis of TTH or migraine according to the International Classification of Headache Disorders (ICHD-II)(1), and expressing voluntary willingness to participate in this study.
  The exclusion criteria for the study included having any pathology involving the cervical region such as disc herniation, radiculopathy, a history of surgery, tumor, or cyst, having received any form of physical therapy targeting the cervical region within the past 3 months, being pregnant or in the menopausal phase; not participating in at least 15% of the training sessions, having a mental disorder (being diagnosed with depression or using antidepressant medication), having a chronic, neurological, or rheumatic disorder; suffering from sinusitis, and being on continuous prophylactic medication for migraines
  Interventions: Other: PROGRESSIVE RELAXATION TRAINING
- WOMEN WITH MIGRAINE (Experimental): The Migraine group consists of 22 women aged 20-45 years.The inclusion criteria were determined as follows being between the ages of 20 and 45, having a diagnosis of TTH or migraine according to the International Classification of Headache Disorders (ICHD-II)(1), and expressing voluntary willingness to participate in this study.
  The exclusion criteria for the study included having any pathology involving the cervical region such as disc herniation, radiculopathy, a history of surgery, tumor, or cyst, having received any form of physical therapy targeting the cervical region within the past 3 months, being pregnant or in the menopausal phase; not participating in at least 15% of the training sessions, having a mental disorder (being diagnosed with depression or using antidepressant medication), having a chronic, neurological, or rheumatic disorder; suffering from sinusitis, and being on continuous prophylactic medication for migraines
  Interventions: Other: PROGRESSIVE RELAXATION TRAINING

INTERVENTIONS:
Other: PROGRESSIVE RELAXATION TRAINING — Both intervention groups were instructed and trained by a physiotherapist 2times a week for 30 minutes each over 6 weeks, The sessions were held in a well-lit, clean and comfortable room with a temperature of 22-24 degrees. Women were asked to stop eating and wear comfortable clothes at least two hours before the sessions. Before the training, relaxation exercises and breathing techniques explained to the women.
  The women lied in the supine position firstly. Then the therapist instructed them to contract and release different muscle groups. They practiced tensing a muscle group until they felt the slight contraction and then released it, simultaneously relaxing other muscle groups. During the session, women were instructed to contract the muscles for 10-20 seconds during deep diaphragmatic breathing and to relax for 30-40 seconds while exhaling.

SUMMARY:
Objective: The aim of this study was to investigate and compare the effects of PRT on pain characteristics, attack frequency, activity self-efficacy perception, and social participation in women with two different types of headaches, TTH and migraine.

Methods: A total of 58 women within the age range of 20 to 45 were screened for eligibility in terms of suitability for participation in the study. Two separate progressive relaxation training sessions were administered to two distinct groups: one comprised of women with TTH and the other consisting of women with migraine. Pre- and post-training assessments were conducted for both groups as follows. Both intervention groups were instructed and trained by a physiotherapist 2times a week for 30 minutes each over 6 weeks,

DETAILED DESCRIPTION:
The International Headache Society (IHS) reported that approximately 90% of headaches consist of tension-type headache (TTH) and migraine, which are the primary type of headache, and affect approximately 50% of the population. The incidence of headaches and migraines is to peak at the age of 20-50, and is more common in women than in men. Recurrent tension-type headaches and migraine attacks negatively affect the quality of life of individuals, reducing working capacity and participation in social and family activities. Therefore, tension-type headaches and migraines cause significant social exclusion, loss of workforce and economic burden.

TTH and migraine impede personal care, productivity and leisure activities, which are an integral part of individuals' lives due to symptoms such as pain, fatigue, difficulty concentrating and/or dizziness. Participation in purposeful activities for individuals is an essential component of health and well-being. Activity self-efficiency is a definition that includes the sense of personal competence and satisfaction about the activities women engage in. When individuals engage in work, play, and daily life activities, women sustain, reinforce, shape, and modify women's capacities, beliefs, and tendencies. High self-efficiency perception can affect the sustainability of physical activity and the productivity of individuals. Both TTH and Migraine tend to occur during the most productive and high-capacity phase of life, between ages 25-55, affecting muscle groups used in daily life activities, potentially leading to limitations in participation, coping, and self-management skills among women. In this regard, it is important to study how tension-type headaches and migraines, which have significant social and individual effects, alter the self-sufficiency and perception of activity in women. Constant thinking of pain and avoiding physical activity can reveal dysfunction in individuals. Because of the individual-specific and complex structure of human roles, each individual suffering from a headache faces different limitations in fulfilling daily roles and social participation, depending on lifestyle and preferences. Thus, non-pharmacological treatments (physiotherapy practices, lifestyle changes, cognitive behavioral therapy, body awareness therapy) are recommended for women with TTH and migraine complaints to relax various muscle groups. One of these treatments is progressive relaxation training. PRT is defined as a method of voluntary, regular relaxation of large muscle groups in the human body with relaxation throughout the body. Specifically, applying PRT to muscle groups found in hands, arms, neck, shoulders, face, chest, abdomen, hips, feet, and fingers, which are most frequently utilized in daily life activities, enhances its benefits for individuals. In the literature, various studies reported that PRT improved occupational performance, participation in daily life activities and quality of life in addition to pain management in individuals with various chronic pains. According to the knowledge, there exists no study in the literature comparing the beneficial effects that PRT, one of the optimal treatments that can be applied in women with TTH or migraine, can have on these two distinct headache groups. Furthermore, studies examining the impact of PRT on activity self-efficacy perception and social participation are quite limited. The aim of this study is to investigate and compare the effects of PRT on pain characteristics, attack frequency, activity self-efficacy perception, and social participation in women with two different types of headaches, TTH and migraine. This study will enable clinicians working with women suffering from TTH and migraine to comprehensively evaluate them in clinical settings and provide more comprehensive intervention approaches to address challenges encountered in daily life.

ELIGIBILITY:
Inclusion Criteria:

* the ages of 20 and 45,
* having a diagnosis of TTH or migraine according to the International Classification of Headache Disorders (ICHD-II)(1), and
* expressing voluntary willingness to participate in this study.

Exclusion Criteria:

* having any pathology involving the cervical region such as disc herniation, radiculopathy, a history of surgery, tumor, or cyst,
* having received any form of physical therapy targeting the cervical region within the past 3 months,
* being pregnant or in the menopausal phase; not participating in at least 15% of the training sessions,
* having a mental disorder (being diagnosed with depression or using antidepressant medication),
* having a chronic, neurological, or rheumatic disorder; suffering from sinusitis, and being on continuous prophylactic medication for migraines

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The incidence of headaches and migraines is to peak at the age of 20-50, and is more common in women than in men (1,2).
Enrollment: 40 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Occupational Self-Assessment (OSA): | up to 5 months
  OSA is a self-reported, client-centered evaluation tool based on MOHO, which assesses the degree of self-awareness and importance of the occupation by measuring the client's ability and value in performing routine occupation. It is a 4-point Likert-type scale consisting of 21 questions and 3 sections.
World Health Organization Disability Assessment Schedule 2 (WHO-DAS II) | up to 5 months
  WHO-DAS II a 36-item general disability instrument that examines difficulties in six domains (activity limitations, communicating ,physical mobility, self-care participation in society, interpersonal interactions, domestic responsibilities and work of life during) in the last 30 days. Responses are given on a 5-point Likert-type scale from 1 (none) to 5 (extreme/cannot do).
Pain Catastrophizing Scale (PCS): | up to 5 months
  The PCS is a 13-item questionnaire comprising three factors, rumination, magnification, and helplessness. Items are scored with a 5-point scale from 0 (not at all) to 4 (all the time). Total score ranges from 0 to 52 (27,28). High scores indicate a high level of catastrophizing.
Headache Impact Test-6: | up to 5 months
  HIT-6, is a 6-item self-administered questionnaire. Items assess headache impact on lost time at work, school or social activities, pain severity, fatigue, frustration, and difficulty with concentration (21,22). Cut scores indicate the following categories: grade 1 (no effect if the scale score is ≤49), grade 2 (50-55 some impact), grade 3 (56-59 substantial impact), grade 4 (≥60 as a severe impact).
Visual Analog Scale (VAS): | up to 5 months
  Pain intensity was assessed with a 10-cm visual analogue scale (VAS). The VAS is scored on a 10- cm horizontal line with indicating 0 'no pain' and 10 'unbearable pain'. The women were asked to mark their headache pain on the horizontal line. (18).

SECONDARY OUTCOMES:
Migraine Disability Assessment Scale (MIDAS): | up to 5 months
  MIDAS is a questionnaire designed to assess disability due to migraine in relation to work, household chores, and family, social or recreational activities over a three-month period (19,20). The MIDAS score is derived from responses reflecting the number of days missed due to headache and the occurrence of days with a 50% reduction in performance

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author, (gkcnakyrk@gmail.com).

REFERENCES:
- [Derived] Karakus A, Uzelpasaci E, Akyurek G. The comparative effectiveness of progressive relaxation training on pain characteristics, attack frequency, activity self-efficacy, and pain-related disability in women with episodic tension-type headache and migraine. PLoS One. 2025 Apr 28;20(4):e0320575. doi: 10.1371/journal.pone.0320575. eCollection 2025. PMID 40293994